CLINICAL TRIAL: NCT05241600
Title: Coping With it All From Labor to Maternity
Brief Title: Neurobehavioral Effects of Prenatal Mindfulness Training on Maternal Presence and Compassionate Love
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidemarie Laurent (Other)
Collaborators: Mind and Life Institute, Hadley, Massachusetts (Other); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor-Investigator, Heidemarie Laurent, Associate Professor of Human Development and Family Studies, Penn State University
Organization: Penn State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19138; 19461 (Other: University of Illinois)
Record Dates: First submitted 2022-01-26; First posted 2022-02-16 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-06

CONDITIONS: Maternal-Fetal Relations; Mother-Child Relations; Maternal Behavior
Keywords: Perinatal; Maternal Mental Health; Mother-Infant Bonding

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either the MBCP condition (intervention under study) or treatment as usual condition (non-mindfulness-based childbirth class of participant's choice from a list provided).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness-Based Childbirth and Parenting (MBCP) (Experimental): Child-bearers randomized to MBCP participate in the 9-week course with a partner (co-parenting partner or other support person who will be involved in the birth). During the training, mothers receive instruction in formal and informal mindfulness practices, and how these apply to the experience of childbirth and parenting an infant. Each weekly 3-hour class includes demonstration and discussion of a practice to be carried out at home over the coming week.
  Interventions: Behavioral: Mindfulness-Based Childbirth and Parenting
- Treatment as Usual (TAU) (Active Comparator): Child-bearers randomized to the treatment as usual comparison group participate (also with a partner) in a non-mindfulness-based childbirth class of their choice from a list provided. To maintain ecological validity of this treatment as usual condition, using an established comparative-effectiveness/pragmatic trial approach, no attempt is made to control the length or contact hours of the class.
  Interventions: Behavioral: Non-Mindfulness-Based Childbirth Class

INTERVENTIONS:
Behavioral: Mindfulness-Based Childbirth and Parenting — MBCP is an adaptation of MBSR that incorporates both standard mindfulness practices (body scan, sitting meditation, mindful movement) and preparation for mindful birthing and parenting an infant. The class is taught by experienced midwives or social workers who have completed MBCP training requirements, which include ongoing cultivation of a personal mindfulness practice as well as education and supervision specific to the MBCP program. See Bardacke (2012) for further description of the MBCP curriculum.
  Arms: Mindfulness-Based Childbirth and Parenting (MBCP)
Behavioral: Non-Mindfulness-Based Childbirth Class — Other childbirth preparation classes available either in-person in the local community or online that do not involve formal mindfulness training will serve as the comparator condition.
  Arms: Treatment as Usual (TAU)

SUMMARY:
This study investigates how prenatal mindfulness training fosters prosocial qualities a mother brings to parenting-specifically, her ability to be present with and experience compassionate love for her child. The mother-child relationship profoundly shapes the way humans learn to experience the world and relate to other people. It is known that mothers who respond more sensitively to their infant's emotional cues form more secure attachment relationships that, in turn, foster positive social-emotional development in the child. Thus, programs that strengthen the capacities supporting maternal sensitivity, such as mothers' ability to attend fully to their child's range of emotions with compassion and lovingkindness, hold great potential for promoting intergenerational well-being. Ideally, such capacities would be cultivated before the child is even born so as to have the greatest cumulative impact.

Mindfulness-Based Childbirth and Parenting (MBCP) is a 9-week program developed to train pregnant women and their partners in the foundations of mindfulness and prepare them to apply mindfulness to birthing and parenting an infant. The intervention has shown beneficial effects on women's psychological wellbeing but has not yet been studied in relation to parenting outcomes. In addition, little is known about (a) biobehavioral mechanisms of action in MBCP, and (b) characteristics of expectant mothers that may moderate the impact of the training. It is important to address these gaps to determine the scope of prenatal mindfulness training effects and who could benefit most from such a program.

This study aims to fill these gaps through an active comparison, randomized controlled trial (RCT) of MBCP compared to (non-mindfulness-based) childbirth education. The investigators will compare mothers who have completed MBCP to mothers with no mindfulness training on both behavioral (self-report) and biological (neural activation to infant cues) indices of prosocial parenting qualities toward the following aims:

Aim 1: Determine the effect of prenatal mindfulness training on self-report measures of maternal presence and compassionate love.

Hypothesis 1: Mothers who have taken part in MBCP will report higher levels of mindful presence, love, and compassion for their infants. These differences will be evident both immediately following the course and sustained later with their infants.

Aim 2: Determine the effect of prenatal mindfulness training on neural activation to one's infant in regions supporting presence and compassionate love.

Including neural measures may reveal intervention effects not yet obvious at the behavioral level that have important consequences for mother/infant functioning.

Hypothesis 2: Mothers who have taken part in MBCP will show increased neural activation to their infant's emotion cues in brain regions involved in present-centered attention (anterior cingulate cortex [ACC] and dorsolateral prefrontal cortex [dlPFC]), emotional resonance (ACC, insula, ventral prefrontal cortex [vPFC]), and mammalian bonding (striatum).

Aim 3: Identify moderating factors that strengthen the effects of prenatal mindfulness training.

Hypothesis 3: Mothers who begin the class with more risk characteristics (single parent, greater distress) will show greater benefits of MBCP, as will those with higher mindfulness practice dosage.

Addressing these aims will shed much-needed light on the ways that mindfulness training during a key developmental life transition can enhance prosocial qualities that contribute to the health and well-being of subsequent generations.

DETAILED DESCRIPTION:
This study was initiated at the PI's previous institution, the University of Illinois at Urbana-Champaign (UIUC), under the approval of the UIUC IRB (protocol 19461). Data collection for participants enrolled at UIUC was concluded in December 2021, and study recruitment and data collection for the remainder of the total sample is to commence at the PI's current institution, the Pennsylvania State University, in January 2022.

Study Procedures

At 20-28 weeks of pregnancy, participants recruited into the study provide informed consent and complete questionnaire measures either in person at the research lab or remotely via phone or Zoom (baseline assessment). Those randomized to MBCP then complete the 9-week class with their partner or other support person, and those assigned to treatment as usual complete an in-person or online birthing class of their choice from a list provided. After taking part in the birthing class, at approximately 37 weeks of pregnancy, women again complete questionnaires remotely (post-class assessment). At 3-4 months postpartum, women complete a final set of questionnaires and take part in a videorecording session with their infant, followed by a brain scanning session at the university-affiliated neuroimaging center.

Consent: Participants who are deemed eligible for the study are contacted to schedule a consent session (in-person or remote). A trained researcher discusses the study protocol and key details of informed consent. Following consent, the researcher discusses what the MRI session will be like and the participant fills out an online safety screener to identify any MRI contraindications. Participants are also asked about availability for birthing classes and to rank the available birthing classes according to their preference.

Birthing Class Assignment + Pre-Class Questionnaire (T1): Between the participant's 20th and 28th week of pregnancy, a study researcher randomly assigns the participant to the treatment (MBCP) or control (birthing class of the participant's choice) condition. The researcher contacts the participant to schedule a birthing class assignment session (T1; by phone or on Zoom). During the birthing class assignment, participants are told whether they have been assigned to the MBCP course or are able to choose a birthing class from the provided list. They are asked whether they have any questions about their assignment and provided with instructions on how to sign up for their class/seek reimbursement, as needed. Following the session, participants are sent a personalized link to the first questionnaire by email for them to complete.

Child-bearers randomized to MBCP complete the 9-week class with their partner or other support person. The class is taught by experienced midwives or social workers who have completed MBCP teacher training requirements, which include ongoing cultivation of a personal mindfulness practice as well as education and supervision specific to the MBCP program. Participants in this condition have the option of participating in one of several online MBCP classes available that accommodates their pregnancy timeline. Each three-hour MBCP class comprises a mix of instructor-guided mindful meditation practice (e.g., engaging in a body scan, breath meditation; prenatal yoga practice) and inquiry, in which instructors lead discussion of participants' experiences of the practice and how it applies to their lives. Classes also involve psychoeducation on the experience of and ways to engage with pregnancy, birth, and parenting from a mindfulness perspective. Participants are encouraged to engage in at-home practice: at least thirty minutes of formal and/or informal mindfulness practices modeled in class six days a week, and to read Mindful Birthing, a companion book written by MBCP developer Nancy Bardacke.

Child-bearers randomized to the treatment as usual group participate (also with a partner) in a childbirth class of their choice from a list provided. To maintain ecological validity of this treatment as usual condition, using an established comparative-effectiveness/pragmatic trial approach, no attempt is made to control the length or contact hours of the class, but a range of classes with varying time commitments are offered, and this information is collected at the post-class assessment and considered as a control variable in analyses. No data collection occurs during any of the classes.

Post-Class Assessment (T2): At approximately 37 weeks of pregnancy (following birthing class completion), participants are emailed a personalized link to a post-class questionnaire for them to complete at home.

Post-Birth Assessment (T3.1): Approximately three months after their infant is born, participants are emailed a personalized link to a post-birth questionnaire for them to complete at home.

Videorecording Visit (T3.2): If the participant indicates they are comfortable with in-person sessions, a researcher schedules a time to visit their home to videorecord the participant interacting with their infant. At the start, mothers are instructed to play with their infant as they normally would for ten minutes (freeplay). Mothers can feel free to play games, sing, use toys, or read books during freeplay. Following freeplay, mother are asked to engage in a structured peekaboo interaction with their infant, which is designed to elicit positive infant affect. During peekaboo, mothers are asked to hold their hands over their eyes and call their baby's name, then reveal their eyes and say "peekaboo." They repeat the above for two and a half minutes. This task may be repeated up to two more times, if needed.

Then mothers are asked to engage in an arm-restraint task (holding the infant's arms gently by their side to restrict movement while adopting a neutral, still expression), a task designed to elicit distress in infants at this age. This task lasts up to two and a half minutes, although the researcher may stop this task early if the baby is quite distressed. Two 12-second video segments each of infant positive and negative emotion expression (4 total) are selected for presentation in the scanner. Positive/negative video segments of an infant not involved in the study are also collected using similar procedures to create the "other infant" stimuli. Non-infant comparison stimuli are created by editing the unfamiliar infant videos using Matlab Image Scramble and time-domain audio scrambling with shufflewins to create scrambled videos with similar audiovisual characteristics but no recognizable infant features.

Brain Scanning Session (T3.3): After the home visit, participants are scheduled for an MRI session at the university-affiliated neuroimaging center. During this session, participants complete five study scans: two resting state scans (6 minutes, 12 seconds each), a structural scan (5 minutes, 21 seconds), and two functional scans where they view the video clips of their own and another unknown infant, as well as non-infant stimulus blocks (8 minutes, 12 seconds each). The total duration of the scan is 45 minutes.

Functional Scanning - Regional brain activity is assessed with blood oxygen level dependent echoplanar images (BOLD-EPI), T2*-weighted gradient echo sequence, TR = 2 s, TE = 25 ms, flip angle = 90 deg, 38 slices of thickness 3.0 mm, with a slice gap of 0.3 mm, 92 x 92 voxel matrix, FOV = 230 mm.

Structural Scanning - Functional data are mapped onto high-resolution T1-weighted structural images using 3-DMagnetization-Prepared RApid Gradient Echo (MPRAGE) pulse sequence, TR = 23000 ms, TE = 2.32 ms, TI = 900 ms, flip angle = 8 deg, 192 sagittal slices of thickness 0.9 mm, 256 x 256 matrix, FOV = 240 mm.

Mothers view the videos via a mirror positioned over their eyes and hear accompanying sounds via headphones (sound check prior to scanning to ensure audibility). Functional runs present each stimulus block 6 times (3 presentations each of unique positive and negative own infant/other infant/scrambled video segments), in counterbalanced order. Video stimuli accompanied by sound were chosen based on previous research showing stronger neural responses to dynamic (as opposed to still) emotion faces, and the investigators' own work showing mindfulness-related effects on mothers' neural response to similar infant videos. Stimulus presentation protocols were informed by previous maternal neuroimaging research. Following scanning, mothers are asked through both open-ended and forced-choice questions what they were doing during the task (distraction or suppression of emotion, mindfulness practice, etc.). They also rate their own and their infant's emotional valence and intensity during each video segment. Reported activities and emotion ratings will be considered as possible covariates in fMRI analysis.

Study Data Analysis

Baseline characteristics of the sample, stratified by experimental group, will be examined to ensure even distribution of key variables. Completers and drop-outs will be compared on baseline variables, and those showing group differences will be considered as covariates in tests of hypotheses. Primary analyses will be conducted with the full sample according to intent-to-treat principles under CONSORT guidelines.

Aim 1: MBCP > self-reported maternal presence and compassionate love. To test Hypothesis 1 that MBCP mothers will show higher levels of these qualities, both following the course and later with their infants, hierarchical linear modeling (HLM) will be used to examine the main effect of experimental group (expressed as a dummy-coded variable indicating MBCP participation) on slopes of self-report measures of presence and compassionate love across all three assessments, as well as post-intervention levels. These models will demonstrate whether MBCP results in increased levels of these qualities, both more generally and specifically with the mother's own infant.

Aim 2: MBCP > neural response to one's infant. To test Hypothesis 2 that MBCP mothers will show increased neural activation to their infant's emotion cues in brain regions supporting the above qualities-i.e., ACC, dlPFC, insula, vPFC, and striatum-group comparisons will be conducted using the FSL program.

At the intrasubject level, multiple regression with OLS and adjustment for autocorrelation will test contrasts of stimulus-specific regressors. Boxcar models reflecting onset-offset of each infant stimulus will be convolved with an optimal basis set for HRF, generated using FLOBS. Results will be averaged across the 2 runs using fixed-effects analysis. Based on both theorized MBCP mechanisms of action and previous research on mindfulness-related maternal brain effects, two aspects of maternal neural response will be examined as outcomes: (1) more general responsiveness to their infant, indexed by contrasts of activation to own > other infant and own-infant > non-infant videos, and (2) valenced responses to their infant, indexed by contrasts of positive > negative own-infant videos.

At the group level, MBCP-related differences in each of these responses will be tested via MBCP > Control and Control > MBCP contrasts with mixed-effects analysis (FLAME) in the whole brain. Cluster threshold correction with Z > 2.6 and FDR < .05 will be used to define regions of significantly different activation, and correspondence with brain atlas-defined anatomical regions will determine whether hypothesized sites of elevated responsiveness are supported.

Aim 3: Identify MBCP moderators. To test Hypothesis 3 that mothers who begin the class with more risk characteristics and/or who receive a higher dosage of mindfulness practice will show greater benefits of MBCP, interaction terms involving moderator variables will be added to the above models. Based on the hypotheses outlined above, investigators expect significant positive interactions between MBCP participation and single relationship status, distress, and practice dosage.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women who

1. Are less than 28 weeks pregnant.
2. Are expecting a singleton child.
3. Are between 18 and 40 years old.
4. Speak English: Because many of the measures employed in the study have not been validated in other languages, we would not be able to offer equivalent birthing classes in other languages, and we do not have researcher staff who are fluent in other languages, participants must be able to understand written/spoken English.
5. Have a Penn State Worry Questionnaire score greater than 50.
6. Live within 40 miles and are willing to come for brain scanning to the university-affiliated neuroimaging center OR live greater than 40 miles away and are willing to travel for the videorecording and brain scanning sessions.

Exclusion Criteria:

Pregnant women/new mothers will be excluded if they have

1. MRI contraindications
2. A serious medical or mental health condition that could impact their ability to participate in study activities. Should a participant endorse a medical or mental health condition that could prevent them from participating in study activities or sessions, a research coordinator, in consultation with the PI, will have a discussion with the participant about whether they feel their condition would prevent them from participating.
3. An existing formal mindfulness or long-term yoga practice

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Five Facet Mindfulness Questionnaire | Time 1 (20-28 weeks pregnancy) through Time 3 (3 months postnatal)
  Measure of maternal mindful presence across time points; score range 1-5; higher scores indicate better outcome.
Inventory of Mindfulness in Parenting - Infant Measure | Time 3 (3 months postnatal)
  Measure of maternal mindful presence with infant at final time point; score range 1-5; higher scores indicate better outcome.
Compassion Scale | Time 1 (20-28 weeks pregnancy) through Time 3 (3 months postnatal)
  Measure of maternal compassion across time points; score range 1-5; higher scores indicate better outcome.
Prenatal Antenatal Attachment Scale | Time 1 (20-28 weeks pregnancy) and Time 2 (37 weeks pregnancy)
  Measure of maternal bonding with fetus at first two time points; score range 1-5; higher scores indicate better outcome.
Maternal Postnatal Attachment Scale | Time 3 (3 months postnatal)
  Measure of maternal bonding with infant at final time point; score range 1-5; higher scores indicate better outcome.
Maternal Neural Response to Infant | Time 3 (3 months postnatal)
  Mothers' BOLD signal during the infant task; functional MRI scans will be analyzed as described above. In particular, two aspects of maternal neural response will be examined as outcomes: (1) more general responsiveness to their infant, indexed by contrasts of activation to own > other infant and own infant > non-infant videos, and (2) valenced responses to their infant, indexed by contrasts of positive > negative own infant videos.

SECONDARY OUTCOMES:
Edinburgh Postnatal Depression Scale | Time 1 (20-28 weeks pregnancy) through Time 3 (3 months postnatal)
  Measure of maternal distress (mood problems) across time points; score range 0-3; higher scores indicate worse outcome.
Perceived Stress Scale | Time 1 (20-28 weeks pregnancy) through Time 3 (3 months postnatal)
  Measure of maternal distress (subjective stress) across time points; score range 0-4; higher scores indicate worse outcome.
Penn State Worry Questionnaire | Time 1 (20-28 weeks pregnancy) through Time 3 (3 months postnatal)
  Measure of maternal distress (anxiety) across time points; score range 1-5; higher scores indicate worse outcome
Center for Epidemiologic Studies Depression Scale | Time 1 (20-28 weeks pregnancy) through Time 3 (3 months postnatal)
  Measure of maternal distress (depression) across time points; score range 0-3; higher scores indicate worse outcome
Ruminative Responses Scale | Time 1 (20-28 weeks pregnancy) through Time 3 (3 months postnatal)
  Measure of maternal distress (rumination) across time points; score range 1-4; higher scores indicate worse outcome
Parenting Stress Index - Short Form | Time 3 (3 months postnatal)
  Measure of maternal parenting stress at final time; score range 1-5; higher scores indicate worse outcome
Self-Compassion Scale | Time 2 (37 weeks pregnancy)
  Measure of maternal self-compassion at post-intervention; score range 1-5; higher scores indicate better outcome
Positive and Negative Affect Scale | Time 3 (3 months postnatal)
  Measure of maternal affect at brain scan session; score range 1-5; higher scores for Positive indicate better outcome; higher scores for Negative indicate worse outcome

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Illinois Urbana-Champaign, Champaign, Illinois
  - Penn State University, University Park, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided
We do plan to share some portion of (deidentified) data in an open access research platform but are still determining which types of data to share and what the most appropriate platform would be.

REFERENCES:
- [Background] Bardacke, N. (2012). Mindful birthing: Training the mind, body, and heart for childbirth and beyond. HarperCollins.
- [Background] Duncan LG, Bardacke N. Mindfulness-Based Childbirth and Parenting Education: Promoting Family Mindfulness During the Perinatal Period. J Child Fam Stud. 2010 Apr;19(2):190-202. doi: 10.1007/s10826-009-9313-7. Epub 2009 Oct 10. PMID 20339571
- [Background] Duncan LG, Cohn MA, Chao MT, Cook JG, Riccobono J, Bardacke N. Benefits of preparing for childbirth with mindfulness training: a randomized controlled trial with active comparison. BMC Pregnancy Childbirth. 2017 May 12;17(1):140. doi: 10.1186/s12884-017-1319-3. PMID 28499376
- [Background] Laurent HK, Ablow JC. The missing link: mothers' neural response to infant cry related to infant attachment behaviors. Infant Behav Dev. 2012 Dec;35(4):761-72. doi: 10.1016/j.infbeh.2012.07.007. Epub 2012 Sep 13. PMID 22982277
- [Background] Laurent HK, Duncan LG, Lightcap A, Khan F. Mindful parenting predicts mothers' and infants' hypothalamic-pituitary-adrenal activity during a dyadic stressor. Dev Psychol. 2017 Mar;53(3):417-424. doi: 10.1037/dev0000258. Epub 2016 Nov 28. PMID 27893234
- [Background] Laurent HK, Wright D, Finnegan M. Mindfulness-related differences in neural response to own infant negative versus positive emotion contexts. Dev Cogn Neurosci. 2018 Apr;30:70-76. doi: 10.1016/j.dcn.2018.01.002. Epub 2018 Jan 5. PMID 29331659
- [Background] Montague DP, Walker-Andrews AS. Peekaboo: a new look at infants' perception of emotion expressions. Dev Psychol. 2001 Nov;37(6):826-38. PMID 11699756
- [Background] Moscardino U, Axia G. Infants' responses to arm restraint at 2 and 6 months: a longitudinal study. Infant Behav Dev. 2006 Jan;29(1):59-69. doi: 10.1016/j.infbeh.2005.07.002. Epub 2005 Aug 3. PMID 17138262
- [Background] Musser ED, Kaiser-Laurent H, Ablow JC. The neural correlates of maternal sensitivity: an fMRI study. Dev Cogn Neurosci. 2012 Oct;2(4):428-36. doi: 10.1016/j.dcn.2012.04.003. Epub 2012 May 10. PMID 22652538
- [Derived] Laurent HK, Haigler KL, Sbrilli MD, Suzuki K, Duncan LG. The relational dimension in mindfulness intervention effects: results of a randomized controlled trial of mindfulness-based childbirth and parenting. BMC Pregnancy Childbirth. 2025 May 10;25(1):560. doi: 10.1186/s12884-025-07676-z. PMID 40348986